CLINICAL TRIAL: NCT02873325
Title: European Patient Registry on Salvage Antiviral Treatment for Patients Experiencing Adenovirus and / or Cytomegalovirus Reactivation Post Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Registry on Salvage Antiviral Treatment for Patients Experiencing ADV and / or CMV Reactivation Post Allogeneic HSCT
Acronym: EPROS
Status: Terminated | Type: Observational
Why Stopped: Lack of study recruitment
Sponsor: Cell Medica Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CM-2016-01
Record Dates: First submitted 2015-10-21; First posted 2016-08-19 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Infectious Complications Following HSCT
Keywords: ADV; CMV; HSCT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: antiviral therapies for CMV and/or ADV — salvage antiviral treatments for ADV and/or CMV

SUMMARY:
DESIGN:

Disease registry - non-interventional.

INDICATION: Patients failing first or subsequent line treatment for adenovirus and / or cytomegalovirus reactivation post allogeneic hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
In this disease registry, data on approximately 120 allo HSCT patients who have received salvage treatment (second or later line) with any antiviral therapy for ADV and / or CMV post allogeneic HSCT will be documented; of these 120, at least 40 patients will have been treated with Cell Medica's immune reconstitution ACT as salvage therapy. The patients will be consented prospectively or retrospectively for collection of data. Data will be collected at baseline, 6 months and 1 year after commencement of salvage treatment. Retrospective data collection (for patients who underwent HSCT in 2010 or later) is permitted.

ELIGIBILITY:
1. Written informed consent
2. Physician requested salvage (defined as refractory to first, requirement for second line or greater) treatment for ADV and / or CMV reactivation post allogeneic HSCT.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this disease registry, data on approximately 120 allo HSCT patients who have received salvage treatment (second or later line) with any antiviral therapy for ADV and/or CMV post allogeneic HSCT will be documented; of these 120, at least 40 patients will have been treated with Cell Medica's immune reconstitution ACT as salvage therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
ADV and/or CMV reactivations | 12 months
  assessment of ADV/CMV viral clearance to evaluate the efficacy of salvage therapies for ADV and / or CMV infections post allogeneic HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Prashant Hiwarkar, Principal Investigator — Birmingham Children's Hospital
Locations (2):
- United Kingdom (2):
  - Birmigham Children Hospital, Birmingham
  - Bristol Royal Hospital For Children, Bristol

IPD SHARING:
Plan to Share IPD: Yes